CLINICAL TRIAL: NCT06892886
Title: Using Immersive Virtual Reality for the Upper Limb Rehabilitation of Post-stroke Subjects: a Multicenter Randomized Control Trial
Brief Title: Using Immersive Virtual Reality for the Upper Limb Rehabilitation of Post-stroke Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Ospedale Accreditato Villa Bellombra (Unknown); Casa di Cura Città di Rovigo (Unknown); IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR_STROKE_MULTICENTER
Record Dates: First submitted 2023-01-30; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Sub-acute Stroke
Keywords: stroke; rehabilitation; upper limb; immersive virtual reality; head-mounted display; subacute stroke
MeSH Terms: conditions — Stroke | interventions — Smart Glasses

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization scheme will be generated using the website http://www.randomization.com and managed by an external administrator. The clinicians who will perform the outcome assessment will be blind regarding the subject's group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): All participants will receive an hour of VR training 5 times/week for 4 weeks within the daily rehab routine.
  Interventions: Device: Virtual Reality
- Control group (No Intervention): Participants will receive the usual rehabilitation activities due to their clinical needs (physical therapy, speech therapy, etc) for 5 times/week over 4 weeks.

INTERVENTIONS:
Device: Virtual Reality — Four tasks, uni and bi-manuals, will be proposed for the treatment of the patient's paretic upper limb in virtual-apartment for improving the relevance and the transferability of the movements requested.
  Other Names: Head-mounted display
  Arms: VR group

SUMMARY:
Stroke produces brain damages that results in sensory, motor, and cognitive impairments which reduce the patient's quality of life and social participation. Upper limb recovery is a complex process whose goal is to allow the patients to gain, in part or completely, independence in daily living activities, for that it represents one of the most important rehabilitation focus. Virtual reality is a fairly recent approach able to simulate concrete movements and functional tasks in a higher dosage compared to other therapies. It seems that the use of VR could improve limb function, however, the amount of this gain is still unclear because of insufficient evidence. This study aims at quantitatively investigating the effectiveness of an HMD immersive virtual reality system on the upper limb functioning in subacute stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of first, ischemic or hemorrhagic, stroke verified by brain imaging within 4 week
* upper limb motor impairment defined by an upper extremity score <55 on the Fugl-Meyer Assessment

Exclusion Criteria:

* neurological conditions in addition to stroke that may affect motor function
* other medical conditions likely to interfere with the ability to safely complete the study protocol
* impaired cognitive functioning that influences the ability to give informed consent
* severe neuropsychological disorders
* visual impairment
* severe upper-limb pain defined as > 7 on the Visual Analogue Scale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in upper limb impairment | Score changes before (T0) and after (T1) the 4 weeks of treatment and at 6-month follow-up (T2)
  Motor recovery will be assessed through the Fugl Meyer Assessment - Upper Extremity

SECONDARY OUTCOMES:
Change in Spasticity | Score changes before (T0) and after (T1) the 4 weeks of treatment and at 6-month follow-up (T2)
  Spasticity grade at the paretic upper limb will be measured with the Ashworth Scale (0-5), in which higher scores are related to more severe muscle hypertonia
Change in Activities of Daily Living | Score changes before (T0) and after (T1) the 4 weeks of treatment and at 6-month follow-up (T2)
  Patient's independence will be quantified with the Barthel Index
Change in perceived quality of life | Score changes before (T0) and after (T1) the 4 weeks of treatment and at 6-month follow-up (T2)
  Stroke Impact Scale 2.0 will be performed for investigating the perceived quality of life, higher scores indicate better quality of life perceived
Kinematic data | Parameters changes (e.g. hand peak velocities) before (T0) and after (T1) the 4 weeks of treatment
  Instrumental data of hand movements registered during the sessions (relevant kinematic indexes will be recorded and offline analyzed such as hand trajectories and peak velocity)
Electroencephalogram | Data changes before (T0) and after (T1) the 4 weeks of treatment (4 weeks) and at 6-month follow-up (T2)
  The EEG signals will be measured by means of a 32-channel cap, according to the International 10-20 system, recorded and monitored by computerized devices.
Treatment satisfaction | After 4 weeks
  The satisfaction related to the virtual training will be investigated through a specific questionnaire
Embodiment | After 4 weeks
  The embodiment feeling will be analyzed with the Gonzalez-Franco questionnaire
Cybersickness | After 4 weeks
  For monitoring undesirable events the Simulator Sickness Questionnaire will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrara University Hospital, Ferrara, Italy